CLINICAL TRIAL: NCT04432558
Title: The Effect of Preoperative Anxiety Level to Postoperative Pain and Analgesic Consumption in Patients Who Had Laparoscopic Sleeve Gastrectomy
Brief Title: Postoperative Effects of Preoperative Anxiety
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yonca Özvardar Pekcan, Medical doctor. Anaesthesia and reanimation specialist, Baskent University
Other Study IDs: K17/24
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Anxiety; Pain, Postoperative
Keywords: Preoperative anxiety level; Postoperative pain; Laparoscopic sleeve gastrectomy
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative | interventions — Tramadol; Acetaminophen; Diclofenac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Preoperative anxiety level
  Interventions: Diagnostic Test: Spielberger's State-Trait Anxiety Inventory
- Postoperative pain and analgesic consumption
  Interventions: Other: Visual analog scale, Ramsay's sedation scale; Drug: Tramadol, paracetamol, diclofenac sodium

INTERVENTIONS:
Diagnostic Test: Spielberger's State-Trait Anxiety Inventory — Patients will be wanted to fill the Spielberger's State-Trait Anxiety Inventory the night before the surgery.
  Groups: Preoperative anxiety level
Other: Visual analog scale, Ramsay's sedation scale — The analgesic consumption of the patients will be recorded by evaluating the pain with VAS (Visual analog scale) and sedation status with Ramsay's sedation scale in the 1st, 4th, 12th and 24th hour of postoperative period.
  Groups: Postoperative pain and analgesic consumption
Drug: Tramadol, paracetamol, diclofenac sodium — The analgesic consumption of the patients will be recorded
  Groups: Postoperative pain and analgesic consumption

SUMMARY:
INTRODUCTION Patients who will have obesity surgery have about %48 psychiatric illnesses like anxiety disorder. Studies which analyze the relationship between preoperative anxiety level and postoperative pain had reported conflicting results. The aim of this study is to search the relationship between preoperative anxiety level and postoperative pain and analgesic consumption in patients who had laparoscopic sleeve gastrectomy surgery.

MATERIAL AND METHODS Our prospective double-blind study is planned to require 86 female patients aged between 18-65 years old, American Society of Anesthesiologists (ASA) I-II and Body mass index (BMI) ≥40 kg/m^2. Patients having a psychiatric or neurologic disease, brain damage, using psychiatric medications (antidepressants, anxiolytics) and chronic alcohol, known allergy to medications used in the study protocol, inability to provide informed consent will be excluded. Patients will be wanted to fill the Spielberger's State-Trait Anxiety Inventory the night before the surgery. The analgesic consumption of the patients will be recorded by evaluating the pain with Visual analog scale (VAS) and sedation status with Ramsay's sedation scale in the 1st, 4th, 12th and 24th hour of postoperative period.

EXPECTATIONS AND SCIENTIFIC CONTRIBUTIONS More satisfying postoperative analgesia may be provided in this group of patients by determining correlation between preoperative anxiety level and postoperative pain and analgesic consumption in patients who had laparoscopic sleeve gastrectomy. Morbidity rate related with pain may be decreased and patient satisfaction may be increased.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18-65 years old
* ASA I-II
* BMI ≥35 kg/m^2

Exclusion Criteria:

* Having a psychiatric or neurologic disease
* Brain damage
* Using psychiatric medications (antidepressants, anxiolytics) and chronic alcohol
* Known allergy to medications used in the study protocol

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients aged between 18-65 years old, ASA I-II, which BMI ≥35 kg/m^2 and have bariatric surgical indications because of morbid (type III) obesity
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Does Preoperative anxiety level effect postoperative pain? | 5 years
  More satisfying postoperative analgesia may be provided in this group of patients by determining correlation between preoperative anxiety level and postoperative pain and analgesic consumption in patients who had laparoscopic sleeve gastrectomy.Patients will be wanted to fill the Spielberger's State-Trait Anxiety Inventory the night before the surgery. The analgesic consumption of the patients will be recorded by evaluating the pain with Visual analog scale (VAS) and sedation status with Ramsay's sedation scale in the 1st, 4th, 12th and 24th hour of postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Zubeyde Hanim Practice and Research Center, Izmir, Karşıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jawaid M, Mushtaq A, Mukhtar S, Khan Z. Preoperative anxiety before elective surgery. Neurosciences (Riyadh). 2007 Apr;12(2):145-8. PMID 21857597
- [Background] Akinsulore A, Owojuyigbe AM, Faponle AF, Fatoye FO. ASSESSMENT OF PREOPERATIVE AND POSTOPERATIVE ANXIETY AMONG ELECTIVE MAJOR SURGERY PATIENTS IN A TERTIARY HOSPITAL IN NIGERIA. Middle East J Anaesthesiol. 2015 Jun;23(2):235-40. PMID 26442401
- [Background] de Zwaan M, Enderle J, Wagner S, Muhlhans B, Ditzen B, Gefeller O, Mitchell JE, Muller A. Anxiety and depression in bariatric surgery patients: a prospective, follow-up study using structured clinical interviews. J Affect Disord. 2011 Sep;133(1-2):61-8. doi: 10.1016/j.jad.2011.03.025. Epub 2011 Apr 17. PMID 21501874
- [Background] Edwards-Hampton SA, Madan A, Wedin S, Borckardt JJ, Crowley N, Byrne KT. A closer look at the nature of anxiety in weight loss surgery candidates. Int J Psychiatry Med. 2014;47(2):105-13. doi: 10.2190/PM.47.2.b. PMID 25084797
- [Background] Clarke H, Kirkham KR, Orser BA, Katznelson R, Mitsakakis N, Ko R, Snyman A, Ma M, Katz J. Gabapentin reduces preoperative anxiety and pain catastrophizing in highly anxious patients prior to major surgery: a blinded randomized placebo-controlled trial. Can J Anaesth. 2013 May;60(5):432-43. doi: 10.1007/s12630-013-9890-1. Epub 2013 Feb 2. PMID 23377862
- [Background] Robleda G, Sillero-Sillero A, Puig T, Gich I, Banos JE. Influence of preoperative emotional state on postoperative pain following orthopedic and trauma surgery. Rev Lat Am Enfermagem. 2014 Oct;22(5):785-91. doi: 10.1590/0104-1169.0118.2481. PMID 25493674
- [Background] Raichle KA, Osborne TL, Jensen MP, Ehde DM, Smith DG, Robinson LR. Preoperative state anxiety, acute postoperative pain, and analgesic use in persons undergoing lower limb amputation. Clin J Pain. 2015 Aug;31(8):699-706. doi: 10.1097/AJP.0000000000000150. PMID 26153780
- [Background] Petrovic NM, Milovanovic DR, Ignjatovic Ristic D, Riznic N, Ristic B, Stepanovic Z. Factors associated with severe postoperative pain in patients with total hip arthroplasty. Acta Orthop Traumatol Turc. 2014;48(6):615-22. doi: 10.3944/AOTT.2014.14.0177. PMID 25637724
- [Background] Ali A, Altun D, Oguz BH, Ilhan M, Demircan F, Koltka K. The effect of preoperative anxiety on postoperative analgesia and anesthesia recovery in patients undergoing laparascopic cholecystectomy. J Anesth. 2014 Apr;28(2):222-7. doi: 10.1007/s00540-013-1712-7. No abstract available. PMID 24077858
- [Background] Aouad MT, Kanazi GE, Malek K, Tamim H, Zahreddine L, Kaddoum RN. Predictors of postoperative pain and analgesic requirements following abdominal hysterectomy: an observational study. J Anesth. 2016 Feb;30(1):72-9. doi: 10.1007/s00540-015-2090-0. Epub 2015 Oct 24. PMID 26499321
- [Background] Bradshaw P, Hariharan S, Chen D. Does preoperative psychological status of patients affect postoperative pain? A prospective study from the Caribbean. Br J Pain. 2016 May;10(2):108-15. doi: 10.1177/2049463716635680. Epub 2016 Mar 2. PMID 27551421
- [Background] De Cosmo G, Congedo E, Lai C, Primieri P, Dottarelli A, Aceto P. Preoperative psychologic and demographic predictors of pain perception and tramadol consumption using intravenous patient-controlled analgesia. Clin J Pain. 2008 Jun;24(5):399-405. doi: 10.1097/AJP.0b013e3181671a08. PMID 18496304
- [Background] Kain ZN, Sevarino F, Alexander GM, Pincus S, Mayes LC. Preoperative anxiety and postoperative pain in women undergoing hysterectomy. A repeated-measures design. J Psychosom Res. 2000 Dec;49(6):417-22. doi: 10.1016/s0022-3999(00)00189-6. PMID 11182434
- [Background] Polomano RC, Heffner SM, Reck DL, Gelnett CM, French D. Evidence for opioid variability, Part 2: Psychosocial influences. Semin Perioper Nurs. 2001 Oct;10(4):159-66. PMID 15129613
- [Background] Caumo W, Hidalgo MP, Schmidt AP, Iwamoto CW, Adamatti LC, Bergmann J, Ferreira MB. Effect of pre-operative anxiolysis on postoperative pain response in patients undergoing total abdominal hysterectomy. Anaesthesia. 2002 Aug;57(8):740-6. doi: 10.1046/j.1365-2044.2002.02690.x. PMID 12133084
- [Background] Ozalp G, Sarioglu R, Tuncel G, Aslan K, Kadiogullari N. Preoperative emotional states in patients with breast cancer and postoperative pain. Acta Anaesthesiol Scand. 2003 Jan;47(1):26-9. doi: 10.1034/j.1399-6576.2003.470105.x. PMID 12492793
- [Background] Feeney SL. The relationship between pain and negative affect in older adults: anxiety as a predictor of pain. J Anxiety Disord. 2004;18(6):733-44. doi: 10.1016/j.janxdis.2001.04.001. PMID 15474849
- [Background] Kalkman JC, Visser K, Moen J, Bonsel JG, Grobbee ED, Moons MKG. Preoperative prediction of severe postoperative pain. Pain. 2003 Oct;105(3):415-423. doi: 10.1016/S0304-3959(03)00252-5. PMID 14527702
- [Background] Hashimoto K, Iwayama S, Sano Y, Tatara T, Hirose M. Preoperative anxiety induces no clinically relevant effect on intraoperative nociceptive levels during breast surgery under general anesthesia. J Anesth. 2015 Dec;29(6):967-70. doi: 10.1007/s00540-015-2032-x. Epub 2015 May 21. PMID 25995061
- [Background] Munafo MR, Stevenson J. Selective processing of threat-related cues in day surgery patients and prediction of post-operative pain. Br J Health Psychol. 2003 Nov;8(Pt 4):439-49. doi: 10.1348/135910703770238293. PMID 14614791
- [Background] Kain ZN, Sevarino FB, Rinder C, Pincus S, Alexander GM, Ivy M, Heninger G. Preoperative anxiolysis and postoperative recovery in women undergoing abdominal hysterectomy. Anesthesiology. 2001 Mar;94(3):415-22. doi: 10.1097/00000542-200103000-00009. PMID 11374599
- [Background] Papageorgiou GM, Papakonstantinou A, Mamplekou E, Terzis I, Melissas J. Pre- and postoperative psychological characteristics in morbidly obese patients. Obes Surg. 2002 Aug;12(4):534-9. doi: 10.1381/096089202762252307. PMID 12194547
- [Background] Kim WS, Byeon GJ, Song BJ, Lee HJ. Availability of preoperative anxiety scale as a predictive factor for hemodynamic changes during induction of anesthesia. Korean J Anesthesiol. 2010 Apr;58(4):328-33. doi: 10.4097/kjae.2010.58.4.328. Epub 2010 Apr 28. PMID 20508787
- [Background] 25. Öner N, Le Compte A. Durumluk-Sürekli Kaygı Envanteri El Kitabı, 1. Baskı, İstanbul, Boğaziçi Üniversitesi Yayınları, 1983; 1-26.
- [Background] Aldrete JA. The post-anesthesia recovery score revisited. J Clin Anesth. 1995 Feb;7(1):89-91. doi: 10.1016/0952-8180(94)00001-k. No abstract available. PMID 7772368
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] 28. Karaman S, Dogru S, Karaman T, Tapar H, Sahin A, Arici S, Kaya Z, Suren M. Anesthesia management in laparoscopic bariatric surgery: Perioperative complications and outcomes in the third year of practice. JCEI 2014; 5: 200-5.
- [Background] Vaughn F, Wichowski H, Bosworth G. Does preoperative anxiety level predict postoperative pain? AORN J. 2007 Mar;85(3):589-604. doi: 10.1016/S0001-2092(07)60130-6. PMID 17352896